CLINICAL TRIAL: NCT04527705
Title: Clinical and Radiographic Outcome of Endodontic Retreatment in One or Two Visits: A Randomized Controlled Trial.
Brief Title: Outcome of Endodontic Retreatment in One or Two Visits
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Juan Gonzalo Olivieri, Principal investigator, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UICENDECL201501
Record Dates: First submitted 2020-08-13; First posted 2020-08-26 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Endodontic Disease; Endodontically Treated Teeth; Root Canal Infection
Keywords: Primary root canal treatment; Secondary root canal treatment; Periapical healing; Outcome
MeSH Terms: conditions — Dental Pulp Diseases; Tooth, Nonvital

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1-vist endodontic retreatment (Active Comparator): Non-surgical root canal retreatment performed in one visit
  Interventions: Procedure: Non-surgical root canal retreatment
- 2-vist endodontic retreatment (Active Comparator): Non-surgical root canal retreatment performed in two visits
  Interventions: Procedure: Non-surgical root canal retreatment

INTERVENTIONS:
Procedure: Non-surgical root canal retreatment — Non-surgical root canal retreatment

SUMMARY:
This study is a prospective randomized controlled study of patients who come to the University and non-surgical root canal retreatment is considered as the election of choice in presence of periapical disease. The aim is to evaluate the success rate of non-surgical retreatment performed in one compared to two visit treatment up to 10 years of follow-up. The null hypothesis is that there will be no statistically significant differences in rates of success, when performing root canal non-surgical retreatment in one or two visits.

ELIGIBILITY:
Inclusion Criteria:

* Patients that demonstrate understanding of the study and willingness to participate as evidenced by signing the voluntary informed consent and received a signed and dated copy of the informed consent form.
* Understands and is willing to comply with all study procedures and restrictions.
* Not presence of clinically significant and relevant abnormalities of clinical history or oral examination.
* Retreatment cases due to an endodontic failure.
* Diagnosis of apical periodontitis.
* Single or bi-radicular teeth.

Exclusion Criteria:

* General: Patients with systemic diseases, diabetes, immunocompromised and pregnant women, or any clinically significant or relevant oral abnormalities.
* Specific: root resorption, root fractures, impossibility of restoration and cases were secondary root canal treatment is not the treatment of choice.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2018-09-20 (Actual); Primary Completion 2021-07-20 (Estimated); Study Completion 2031-07-20 (Estimated)

PRIMARY OUTCOMES:
Clinical post-operative pain | Immediately post treatment
  VAS score (0-10) of patient' level of pain, from no pain to extreme pain
Clinical post-operative pain | 4 hours post-treatment
  VAS score (0-10) of patient' level of pain, from no pain to extreme pain
Clinical post-operative pain | 24 hours post treatment
  VAS score (0-10) of patient' level of pain, from no pain to extreme pain
Clinical post-operative pain | 48 hours post treatment
  VAS score (0-10) of patient' level of pain, from no pain to extreme pain
Clinical signs or symptoms of periapical disease 1 | 1 year
  Absence/presence of clinical signs or symptoms of periapical disease
Clinical signs or symptoms of periapical disease 2 | 2 years
  Absence/presence of clinical signs or symptoms of periapical disease
Clinical signs or symptoms of periapical disease 4 | 4 years
  Absence/presence of clinical signs or symptoms of periapical disease
Clinical signs or symptoms of periapical disease 6 | 6 years
  Absence/presence of clinical signs or symptoms of periapical disease
Clinical signs or symptoms of periapical disease 10 | 10 years
  Absence/presence of clinical signs or symptoms of periapical disease
Radiographic periapical absence/presence of radiographic apical periodontitis | 1 year
  Absence/presence of radiographic apical periodontitis + PAI changes when compared with post-treatment radiograph
Radiographic periapical absence/presence/changes in radiographic apical periodontitis | 2 years
  Absence/presence of radiographic apical periodontitis + PAI changes when compared with post-treatment radiograph
Radiographic periapical absence/presence/changes in radiographic apical periodontitis | 4 years
  Absence/presence of radiographic apical periodontitis + PAI changes when compared with post-treatment radiograph
Radiographic periapical absence/presence/changes in radiographic apical periodontitis | 6 years
  Absence/presence of radiographic apical periodontitis + PAI changes when compared with post-treatment radiograph
Radiographic periapical absence/presence/changes in radiographic apical periodontitis | 10 years
  Absence/presence of radiographic apical periodontitis + PAI changes when compared with post-treatment radiograph

SECONDARY OUTCOMES:
Correlation of prognostic factors and clinical signs or symptoms of periapical disease 1 | 1 year
  Correlation of pre-treatment symptomatology, post-operative pain, radiographic periapical lesion size, being an abutment, and presence of antagonist, in relation to having clinical signs or symptoms of periapical disease
Correlation of prognostic factors and clinical signs or symptoms of periapical disease 2 | 2 years
  Correlation of pre-treatment symptomatology, post-operative pain, radiographic periapical lesion size, being an abutment, and presence of antagonist, in relation to having clinical signs or symptoms of periapical disease
Correlation of prognostic factors and clinical signs or symptoms of periapical disease 4 | 4 years
  Correlation of pre-treatment symptomatology, post-operative pain, radiographic periapical lesion size, being an abutment, and presence of antagonist, in relation to having clinical signs or symptoms of periapical disease
Correlation of prognostic factors and clinical signs or symptoms of periapical disease 6 | 6 years
  Correlation of pre-treatment symptomatology, post-operative pain, radiographic periapical lesion size, being an abutment, and presence of antagonist, in relation to having clinical signs or symptoms of periapical disease
Correlation of prognostic factors and clinical signs or symptoms of periapical disease 10 | 10 years
  Correlation of pre-treatment symptomatology, post-operative pain, radiographic periapical lesion size, being an abutment, and presence of antagonist, in relation to having clinical signs or symptoms of periapical disease

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No